CLINICAL TRIAL: NCT01740050
Title: Effect of Different Weight-loss Methods on Gut-brain Interactions
Brief Title: Weight-loss and Gut-brain Interactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL42676.068.12
Record Dates: First submitted 2012-11-21; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Roux- and Y bypas surgery (RYGB) (Active Comparator): One subject group will lose 10% of initial body weight using RYGB. RYGB is an operation that first divides the stomach into a small upper pouch and a much larger lower "remnant" pouch and then re-arranges the small intestine to connect to both, in this way bypassing part of the small intestine.
  Interventions: Procedure: RYGB
- Laparoscopic adjustable gastric banding (LAGB) (Active Comparator): One subject group will lose 10% of initial body weight using LAGB. With LAGB an inflatable band is placed around the upper part of the stomach to create a smaller stomach pouch. This slows and limits the amount of food that can be consumed at one time giving the opportunity for the sense of satiety to be met. It does not decrease gastric emptying time.
  Interventions: Procedure: LAGB
- Very Low Calorie Diet (VLCD) (Active Comparator): One subject group will lose 10% of initial body weight using a VLCD. There are no risks for the subjects in consuming the VLCD (Modifast, together with the recommended fruit and vegetables) as the macronutrient composition and vitamins/minerals content meet the Dutch recommended daily allowance.
  Interventions: Dietary Supplement: Very Low Calorie Diet (VLCD)

INTERVENTIONS:
Dietary Supplement: Very Low Calorie Diet (VLCD) — One subject group will lose 10% of initial body weight using a VLCD. There are no risks for the subjects in consuming the VLCD (Modifast, together with the recommended fruit and vegetables) as the macronutrient composition and vitamins/minerals content meet the Dutch recommended daily allowance.
  Arms: Very Low Calorie Diet (VLCD)
Procedure: RYGB
  Arms: Roux- and Y bypas surgery (RYGB)
Procedure: LAGB
  Arms: Laparoscopic adjustable gastric banding (LAGB)

SUMMARY:
While exposure to an obesogenic environment has increased for almost every individual in western society, not everyone is equally susceptible to overeating and not everyone becomes obese. Teasing apart the physiological underpinnings of those individual seemingly protective- differences may contribute to the development of successful preventive measures and treatment. Neuroimaging studies started to deliver important insights into the neuroanatomical determination of individual eating behavior. However, food intake is not only determined by the brain, but is orchestrated by an interaction of peripheral hormones with neural circuits and decision-making processes. This interactive axis is also referred to as the gut-brain axis. While individual aspects of the axis have been studied extensively, detailed insight in the interaction of gut and brain in the regulation of food intake is lacking.

Objective: The current study aims to investigate the effect of a) caloric restriction (very low calorie diet (VLCD)); b) caloric restriction with mechanical restriction (Laparoscopic adjustable gastric banding (LAGB)); and c) caloric restriction with mechanical restriction and physiological changes through malapsorption (Roux- en- Y bypass (RYGB) surgery) on gut-brain interactions to find an optimal balance for weight loss and long-term sustained weight maintenance.

DETAILED DESCRIPTION:
Rationale: While exposure to an obesogenic environment has increased for almost every individual in western society, not everyone is equally susceptible to overeating and not everyone becomes obese. Teasing apart the physiological underpinnings of those individual seemingly protective- differences may contribute to the development of successful preventive measures and treatment. Neuroimaging studies started to deliver important insights into the neuroanatomical determination of individual eating behavior. However, food intake is not only determined by the brain, but is orchestrated by an interaction of peripheral hormones with neural circuits and decision-making processes. This interactive axis is also referred to as the gut-brain axis. While individual aspects of the axis have been studied extensively, detailed insight in the interaction of gut and brain in the regulation of food intake is lacking.

Objective: The current study aims to investigate the effect of a) caloric restriction (very low calorie diet (VLCD)); b) caloric restriction with mechanical restriction (Laparoscopic adjustable gastric banding (LAGB)); and c) caloric restriction with mechanical restriction and physiological changes through malapsorption (Roux- en- Y bypass (RYGB) surgery) on gut-brain interactions to find an optimal balance for weight loss and long-term sustained weight maintenance.

Study design: In a repeated measures design a total of 45 obese (body mass index (BMI) > 35 ≤ 45) study participants will be investigated. All participants will undergo a weight loss period of 10% of initial body weight by means of VLCD intervention (n=15), RYGB surgery (n=15) or LAGB surgery (n=15).

Study population: The study population is composed out of people qualifying for a surgical weight loss procedure (RYGB or LAGB). A total of 45 obese (BMI > 35 ≤ 45) study participants between age 18 and 60 will be investigated Intervention: One subject group (n=15) will undergo a diet intervention, which consists of a very low calorie diet (VLCD; Modifast) containing 2.1MJ/d for 1 to 2 months, until they lost 10% of their initial body weight.

This intervention will be compared with 2 other weight loss groups; one group will undergo RYGB surgery and one group will undergo LAGB surgery. However, these surgical procedures will proceed as planned and according to the standard clinical practice, and will in no way be changed.

Main study parameters/endpoints: To determine the optimal interaction of gut hormones and brain activity for successful weight loss and sustained weight maintenance this study will examine the effect of interaction of gastrointestinal hormone release on neural network activation through a) caloric restriction; b) caloric restriction with physiological restriction; and c) caloric restriction with malapsorption on food reward processing and decision making in the brain as well as on gastrointestinal hormone release.

* The main parameters contributing to efficient, effective and satisfactorily weight maintenance at the same time is the change in satiety and in food reward upon an iso-energetic test-meal. This will be the main factor contributing to compliance and preventing reversal, (measured by visual analog scales (VAS), changes in ad libitum meal intake, representation in the brain of food reward processing and decision making, computer test, TFEQ for cognitive restraint, disinhibition and hunger).
* Secondary contributions to this main parameter are:

  * Possible changes in the gut-microbiota population, interacting with neuronal signaling for satiety and reward;
  * The weight loss itself, changes in body-composition, and changes in resting- and diet-induced energy expenditure, all underscoring weight maintenance.
  * Possible changes in the endocannabinoid profile, interacting with neuronal signaling for satiety and reward Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This research is beneficial to the subjects, in that they all, being obese, will loose body-weight. Subjects included in the diet induced weight loss group will lose 10% of their initial weight, which is beneficial for the operation, as it will decrease the risk. This will however not compromise their possibility to undergo surgery if their BMI decreases below 35, as the intake for surgery is based upon the initial screening, proving that they are not able to be weight stable and that they already tried to be at a healthy stable weight with other weight loss methods. All participants will have to come visit the metabolic research unit Maastricht (MURM) on 4 different occasions, twice before the weight loss procedure and twice after. These visits will be combined with regular hospital visits as much as possible.

FMRI is a non-invasive standard method for to determine blood oxygenation in areas of interest without any significant risks (See document section K6 for standardized and approved methods for conducting fMRI experiments involving human subjects). It is a technique that utilizes magnetic fields and low-energy radio frequencies to visualize brain structures and brain function. Through careful screening procedures subjects with metallic fragments in their body will be excluded from the study since the fMRI magnet exerts a force on ferromagnetic objects. During test day 2 (before and after the weight loss procedure) a canula will be inserted for blood sampling. Blood sampling in this study does not include any other risks for the subjects, other than its usual risk of minor bruising.

One subject group will lose 10% of initial body weight using a VLCD. There are no risks for the subjects in consuming the VLCD (Modifast, together with the recommended fruit and vegetables) as the macronutrient composition and vitamins/minerals content meet the Dutch recommended daily allowance. This VLCD will demand some energy from the subjects at home. However, due to extensive experience with VLCD in our laboratory and due to the benefit of weight loss for the participants we anticipate enough will-power to complete these 2 months VLCD.

This intervention will be compared with 2 other weight loss groups; one group will undergo RYGB surgery and one group will undergo LAGB surgery. RYGB is an operation that first divides the stomach into a small upper pouch and a much larger lower "remnant" pouch and then re-arranges the small intestine to connect to both, in this way bypassing part of the small intestine. With LAGB an inflatable band is placed around the upper part of the stomach to create a smaller stomach pouch. This slows and limits the amount of food that can be consumed at one time giving the opportunity for the sense of satiety to be met. It does not decrease gastric emptying time. However, both surgical procedures will proceed as planned and will in no way be changed. Therefore, further explanation is beyond the scope of this protocol.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, a subject must qualify for weight loss surgery with LAGB or RYGB, as evaluated by a physician at intake for surgery. Furthermore, subjects must meet all of the following criteria:

* Subject, male or female, is age 18 to 60 years of age.
* Subject must be able to understand and be willing to sign an informed consent document.
* Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study.
* Subject has a body mass index (BMI) of 40 - 45 or 35 to 39.9 plus one or more co-morbid diseases expected to improve with weight loss, including but not limited to hypertension, dyslipidemia, obstructive sleep apnea, or diabetes mellitus.
* Subject must be of sufficient and stable medical health, as evaluated by physician at intake.
* Subject must have failed standard obesity therapy of diet, exercise, behaviour modification, and pharmacologic agents either alone or in combination, as assessed at the intake for surgery by a physician.
* For the fMRI measurements inclusion criteria are as follows: not having any metallic fragments in the body, being right-handed. Because of the different brain laterality in left- and right-handed subjects we chose to include only right-handed subjects. Hence the results can be compared between the subjects.

Exclusion Criteria:

* - Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease, as evaluated by physician at intake for the surgery.
* Subject has had significant weight loss in the last 3 months (>5kg).
* Subject has a history or is diagnosed with eating disorders.
* Subject has renal and/or hepatic insufficiency, as evaluated by physician at intake.
* Subject has thyroid disease, which is not controlled with medication, as evaluated by physician at intake for the surgery.
* Female subject who is pregnant (i.e., has a positive urine or blood pregnancy test prior to the procedure), is suspected to be pregnant, is lactating or is of childbearing potential but refuses to use adequate contraception during the study.
* Female subject who started birth control pills less than 3 months before enrollment, or who plans to start taking birth control pills during the study.
* Subjects who cannot discontinue either prescription or over the counter weight loss medications for at least 30 days prior to the start of the study as well as during the trial period.
* Subjects who have started medications within the last 3 months that are known to cause weight gain.
* Subjects who have cardiac pacemakers or other electronic implantable devices.
* Subjects who have psychiatric disease including but not limited to manic-depressive disorder, schizophrenia, borderline personality disorder, depression or suicidal tendencies.
* Subject currently uses or has a history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
* Subject has participated in a clinical study with an investigational new drug, biological, or therapeutic device within ≤ 28 days prior to enrollment in this study, and does not agree to abstain from participation in other clinical trials of any kind during this study.
* Presence of contra-indications for f-MRI, as mentioned in the screening form and informed consent of the faculty of psychology (see section E2 and F1).
* Claustrophobia
* Being left-handed
* Metallic fragments in the body

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
the optimal interaction of gut hormones and brain activity | 30 to 60 days: At baseline and after weight loss (10% of initial weight)
  To determine the optimal interaction of gut hormones and brain activity, resulting in successful weight loss and sustained weight maintenance. This objective will be investigated by examining the effect of a) caloric restriction (VLCD); b) caloric restriction with mechanical restriction (LAGB); and c) caloric restriction with mechanical restriction and physiological changes through malapsorption (RYGB) on food reward processing and decision-making in the brain and on gastrointestinal hormone release.
  The main parameters contributing to efficient, effective and satisfactorily weight maintenance at the same time is the change in satiety and in food reward upon an iso-energetic test-meal. This will be the main factor contributing to compliance and preventing reversal, (measured by visual analog scales (VAS), changes in ad libitum meal intake, representation in the brain of food reward processing and decision making, computer test, TFEQ for cognitive restraint, disinhibition and hunger).

SECONDARY OUTCOMES:
gut-microbiota | 30 to 60 days: At baseline and after weight loss (10% of initial weight)
  Possible changes in the gut-microbiota population, interacting with neuronal signaling for satiety and reward;
body composition | 30 to 60 days: At baseline and after weight loss (10% of initial weight)
  The weight loss itself and changes in body-composition; underscoring weight maintenance.
endocannabinoid profile | 30 to 60 days: At baseline and after weight loss (10% of initial weight)
  Possible changes in the endocannabinoid profile, interacting with neuronal signaling for satiety and reward
Diet induced energy expenditure | 30 to 60 days: At baseline and after weight loss (10% of initial weight)
  Changes in resting- and diet-induced energy expenditure; underscoring weight maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja C Adam, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University (metabolic research unit Maastricht (MRUM)), Maastricht, Netherlands